CLINICAL TRIAL: NCT02844478
Title: Effect of Stress-Busting Program on Caregivers' Quality of Life, Stress/Immunity Bio-markers, and Cellular Aging
Brief Title: Stress-Busting Program and QoL, Bio-markers of Immunity/Stress and Cellular Aging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: WellMed Charitable Foundation (Unknown); The Claude D. Pepper Older Americans Independence Centers (Other); The Sam and Ann Barshop Institute for Longevity and Aging Studies (Unknown); San Antonio Geriatrics Research Education and Clinical Center- GRECC (Unknown); Caring Companions (Unknown); Alzheimer's Association (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HSC20160309H
Record Dates: First submitted 2016-07-20; First posted 2016-07-26 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Stress, Psychological; Telomere Shortening; Stress, Physiological
Keywords: Caregiving; Family caregiving; Stress; dementia caregiving; Hispanics; Spanish; Telomere
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SBP ENGLISH (Active Comparator): Caregivers will complete the 9 -week Stress-Busting Program for Family Caregivers in English
  Interventions: Behavioral: SBP English
- SBP SPANISH (Experimental): Caregivers will complete the 9 -week Stress-Busting Program for Family Caregivers in Spanish
  Interventions: Behavioral: SBP SPANISH

INTERVENTIONS:
Behavioral: SBP English — The SBP caregiver intervention has been successfully delivered and disseminated in the US. It is currently offered in 9 states and 16 Texas counties . The SBP is designed to a) improve the QoL of family caregivers who provide care for people with ADRD and b) help caregivers manage their stress and cope better with their lives. The SBP is implemented using a Master Trainer/Group Facilitator (lay leader) model. The SBP is a multi-component intervention that meets for 90 minutes once a week for 9 consecutive weeks.
  Other Names: SBP-E
  Arms: SBP ENGLISH
Behavioral: SBP SPANISH — The SBP caregiver intervention has been successfully delivered and disseminated in the US. It is currently offered in 9 states and 16 Texas counties . The SBP is designed to a) improve the QoL of family caregivers who provide care for people with ADRD and b) help caregivers manage their stress and cope better with their lives. The SBP is implemented using a Master Trainer/Group Facilitator (lay leader) model. The SBP is a multi-component intervention that meets for 90 minutes once a week for 9 consecutive weeks. The Spanish translation and cultural adaptation of the SBP has been completed under the direction of the PI.
  Other Names: SBP-S
  Arms: SBP SPANISH

SUMMARY:
The purpose of this study is to explore the differences in quality of life , inflammation, stress, telomere length, and mucosal immune function of Hispanic and non-Hispanic caregivers of persons with Alzheimer's disease and related dementias (ADRD). The caregivers will complete the Stress-Busting Program for Family Caregivers in the language of their choice (English or Spanish).

DETAILED DESCRIPTION:
The overarching goal of this project is to (1) explore the differences in quality of life (QoL), inflammation, stress, telomere length, and mucosal immune function of Hispanic caregivers of persons with ADRD and (2) determine whether a caregiver intervention can effectively improve the QoL, inflammation, stress, telomere length, and mucosal immune function biomarkers of Hispanic caregivers.

The proposed study is a non-randomized trial design with three groups of ADRD caregivers that vary based on Hispanic ethnicity and English/Spanish language preference. The project's specific aims are:

Specific Aim 1: To compare the quality of life (QoL) (stress, depression, and burden), mucosal immunity function (sIgA), stress (sCortisol and sAmylase), inflammation(CRP), and telomere length in Spanish-speaking Hispanic, English-speaking Hispanic, and English-speaking non-Hispanic caregivers who participate in an evidence-based Stress-Busting Program (SBP) for family caregivers of family members living with ADRD. Working hypothesis: At baseline, Spanish-speaking Hispanic caregivers have lower QoL and immune function, higher levels of inflammation and stress, and shorter telomeres as compared to Hispanic and non-Hispanic English-speaking caregivers.

Specific Aim 2: To compare the impact of the SBP on QoL and biomarkers for stress, aging, inflammation and mucosal immunity among those caregivers completing the SBP (Hispanic caregivers completing the culturally adapted translated version to Spanish of SBP and Hispanic and non-Hispanic caregivers completing the English-SBP). Working Hypothesis: Spanish-speaking Hispanic caregivers completing the Spanish-SBP show more improvement in their QoL and biomarkers of stress, mucosal immunity, aging and inflammation post-intervention as compared to Hispanic and Non-Hispanic caregivers completing the English-SBP. To achieve these aims, the investigators propose to deliver the 9-week English SBP and the translated and culturally adapted Spanish-SBP. Saliva and blood samples and self- report measures of QoL will be collected at baseline and 9 weeks (end of intervention)

ELIGIBILITY:
Inclusion Criteria:

1. self-identified caregiver for a person living with ADRD. Family caregivers of people with ADRD include spouses, adult children, grandchildren, siblings, partners, and significant others.

   In addition to Alzheimer's disease, other causes of dementia include multiple sclerosis, Parkinson's, post-traumatic stress disorder (PTSD), and/or traumatic brain injury (TBI),
2. over the age of 18,
3. those wishing to participate in the Spanish SBP must speak and read Spanish.

Exclusion Criteria:

* Speaking a language other than English or Spanish
* Caring for an individual not diagnosed with a cognitive impairment as delineated in inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Telomere length | Baseline and end of intervention (Week 9)

SECONDARY OUTCOMES:
Salivary flow rate | Baseline and end of intervention (Week 9)
Saliva potential hydrogen (pH) | Baseline and end of intervention (Week 9)
Salivary protein | Baseline and end of intervention (Week 9)
Perceived Stress Scale | Baseline and end of intervention (Week 9)
Center for Epidemiologic Depression (CES-D) | Baseline and end of intervention (Week 9)
Screen for Caregiver Burden | Baseline and end of intervention (Week 9)
Salivary alpha Amylase (sAA) | Baseline and end of intervention (Week 9)
Secretory immunoglobulin A (SIgA) | Baseline and end of intervention (Week 9)
C Reactive Protein (CRP) | Baseline and end of intervention (Week 9)

CONTACTS AND LOCATIONS:
Overall Officials: Lyda C Arevalo-Flechas, PhD, RN, Principal Investigator — Audie L. Murphy VA Hospital, STVHCS; Chih-Ko Yeh, BDS, PhD, Principal Investigator — Audie L. Murphy VA Hospital, STVHCS
Locations (1):
- The University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lewis SL, Miner-Williams D, Novian A, Escamilla MI, Blackwell PH, Kretzschmar JH, Arevalo-Flechas LC, Bonner PN. A stress-busting program for family caregivers. Rehabil Nurs. 2009 Jul-Aug;34(4):151-9. doi: 10.1002/j.2048-7940.2009.tb00271.x. PMID 19583056
- [Background] Lucke KT, Martinez H, Mendez TB, Arevalo-Flechas LC. Resolving to go forward: the experience of Latino/Hispanic family caregivers. Qual Health Res. 2013 Feb;23(2):218-30. doi: 10.1177/1049732312468062. PMID 23258419
- [Background] Arevalo-Flechas LC, Acton G, Escamilla M, Bonner P, Lewis SL. Latino Alzheimer's caregivers: What is important to them?. Journal of Managerial Psychology. 2014; 6(29):661-684
- [Background] Arevalo-Flechas LC. Beyond translated consents: Culturally competent research. Perioperative Nursing Clinics. 2009; 4(3):287 - 296.
- [Background] Medrano MA, DeVoe PH, Padilla A, Arévalo-Flechas LC. A targeted review to examine reporting of translation methodology in Hispanic health studies. Hispanic health care international : the official journal of the National Association of Hispanic Nurses. 2010; 8(3):145 - 153
- [Background] Arévalo-Flechas LC, Lewis SL. Lost in translation: What does burden mean to Latino caregivers? [Abstract]. Journal of the American Geriatrics Society. 2006;54(4):S177
- [Background] Turner RM, Hinton L, Gallagher-Thompson D, Tzuang M, Tran C, Valle R. Using an Emic lens to understand how Latino families cope with dementia behavioral problems. Am J Alzheimers Dis Other Demen. 2015 Aug;30(5):454-62. doi: 10.1177/1533317514566115. Epub 2015 Jan 19. PMID 25601209
- [Background] Hinton L, Haan M, Geller S, Mungas D. Neuropsychiatric symptoms in Latino elders with dementia or cognitive impairment without dementia and factors that modify their association with caregiver depression. Gerontologist. 2003 Oct;43(5):669-77. doi: 10.1093/geront/43.5.669. PMID 14570963
- [Background] Ortiz F, Fitten LJ, Cummings JL, Hwang S, Fonseca M. Neuropsychiatric and behavioral symptoms in a community sample of Hispanics with Alzheimer's disease. Am J Alzheimers Dis Other Demen. 2006 Aug-Sep;21(4):263-73. doi: 10.1177/1533317506289350. PMID 16948291
- [Background] Gallagher-Thompson D, Coon DW, Solano N, Ambler C, Rabinowitz Y, Thompson LW. Change in indices of distress among Latino and Anglo female caregivers of elderly relatives with dementia: site-specific results from the REACH national collaborative study. Gerontologist. 2003 Aug;43(4):580-91. doi: 10.1093/geront/43.4.580. PMID 12937336
- [Background] Vitaliano PP, Russo J, Young HM, Becker J, Maiuro RD. The screen for caregiver burden. Gerontologist. 1991 Feb;31(1):76-83. doi: 10.1093/geront/31.1.76. PMID 2007478
- [Background] Radloff LS.The CES-D Scale: A self-report depression scale for research in the general population. Applied Psychological Measurement. 1977;1:385-408.
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Piazza JR, Almeida DM, Dmitrieva NO, Klein LC. Frontiers in the use of biomarkers of health in research on stress and aging. J Gerontol B Psychol Sci Soc Sci. 2010 Sep;65(5):513-25. doi: 10.1093/geronb/gbq049. Epub 2010 Jul 20. PMID 20647348
- [Background] Granger DA, Kivlighan KT, el-Sheikh M, Gordis EB, Stroud LR. Salivary alpha-amylase in biobehavioral research: recent developments and applications. Ann N Y Acad Sci. 2007 Mar;1098:122-44. doi: 10.1196/annals.1384.008. Epub 2007 Mar 1. PMID 17332070
- [Background] Yeh CK, Johnson DA, Dodds MW. Impact of aging on human salivary gland function: a community-based study. Aging (Milano). 1998 Oct;10(5):421-8. doi: 10.1007/BF03339889. PMID 9932146
- [Background] Arévalo-Flechas LC. Factors influencing Latino/Hispanic caregivers' perception of the experience of caring for a relative with Alzheimer's disease. Dissertation Abstracts International. DAI-B 69/066
- See also: Pew Research Center statistics on Hispanics. — http://www.pewresearch.org/fact-tank/2014/12/16/with-fewer-new-arrivals-census-lowers-hispanic-
- See also: Technology Engineering and Design (TEDx) presentation: All Alzheimer's Caregivers are not Created Equal. — https://youtu.be/2QYdXGZNp5A
- See also: Factors influencing Hispanic caregivers' perception of the experience of caring for a relative with Alzheimer's disease — http://pqdtopen.proquest.com/pubnum/3311328.html